CLINICAL TRIAL: NCT03488888
Title: Evaluation of Pectoral Nerve Blocks II for Augmentation Mammoplasty Surgeries. Prospective, Randomized, Double-blind Study
Brief Title: PEC Block II in Mammoplasty Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Leonardo Henrique Cunha Ferraro, Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEC Block
Record Dates: First submitted 2017-07-14; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Mammaplasty; Anesthesia, Conduction; Analgesia; Analgesia, Patient-Controlled
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal Saline (Sham Comparator): General Anesthesia + Bilateral Pectoral injection of Normal Saline 0,9%
  1. Ultrasound-guided visualization of Pectoralis major and pectoralis minor muscles
  2. Injection of 10 mL normal saline 0,9% between muscles lateral to the thoracoacromial artery.
  3. Visualization of Pectoralis menor and Serratil Muscles
  3- Injection of 20 mL of normal saline 0,9% between Pectoralis minor and serratil muscles 4-Visualize the hydrodissection performed by the solution
  Interventions: Drug: Normal Saline 0,9%
- Bupivacaine (Experimental): General Anesthesia + Bilateral Pectoral injection of 30 mL of 0.25% Bupivacaine
  1. Ultrasound-guided visualization of Pectoralis major and pectoralis minor muscles
  2. Injection of 10 mL of local anesthetic between muscles lateral to the thoracoacromial artery.
  3. Visualization of Pectoralis minor and Serratil Muscles
  3- Injection of 20 mL of local anesthestic between Pectoralis minor and Serratil muscles 4-Visualize the hydrodissection performed by the solution
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Normal Saline 0,9% — Ultrasound-guided PEC II block with 30 mL of Normal Saline 0,9%
  Arms: Normal Saline
Drug: Bupivacaine — Ultrasound-Guided PEC block with 30 mL of 0.25% bupivacaine solution
  Other Names: Brand: Cristália
  Arms: Bupivacaine

SUMMARY:
Breast augmentation surgery is the top cosmetic surgery in USA with more then 300.000 cases performed annually. Pain is a common complications of the procedure accompanied of dyspnea and nausea due to the surgical manipulation.

Several anesthetic techniques were developed with the objective of providing optimal surgical conditions together with enhanced recovery and post-op pain management.

Pectoralis major block was first described in 2011 by Blanco in female patients undergoing oncologic procedures in the anterior thoracic wall.

The investigators hypothesized if the Pectoralis Major block combined with general anesthesia standard techniques could be beneficial in improving pain scores and opioid consumption during post operative period of patients undergoing breast augmentation surgery.

DETAILED DESCRIPTION:
Patients undergoing Breast Augmentation Mammoplasty were submitted to laryngeal mask placement after anesthetic induction with Fentanyl 3ucg/kg , Propofol 2mg/kg and Atracurium 0,5mg/kg and surgery was performed under standard surgical practices.

Before the surgical incision patients were randomized either to receive a Bilateral Pectoralis Major Block(PEC I and II) with Bupivacaine 0,25% with Epinephrine or to receive a placebo block with Normal Saline 0,9%.

After the procedure all patients received a intravenous patient-controlled-analgesia pump device with morphine.

Pain and opioid consumption were assessed with a pain score assessment tool and assessment of the pump administration dosage history.

No NSAIDs or alpha 2 agonist drugs were administered during or after the procedure.

The maintenance of anesthesia was performed with Propofol and Remifentanil Total intravenous anesthesia(TIVA) models in a standardized fashion. Micromanagement of anesthetic drugs was performed by the assistant anesthesiologist physician.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Above 18 years old
* Elective Surgery
* American Society of Anesthesia(ASA) Class I up to III

Exclusion Criteria:

* Pregnancy
* Acute Coronary Syndrome
* History of Arrhythmia
* Functional Class New York Heart Association(NYHA) III or IV
* Previous thoracic/breast surgery
* History of Chronic Pain
* Neuromuscular disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-11-03 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Pain Score | 24 hours after surgery
  Patients will be actively questioned about their pain score assessment

SECONDARY OUTCOMES:
Opioid Consumption | 1 hour, 2 hours, 4 hours, 6 hours, 12 hours and 24 hours after surgery
  The total amount of opioid will be evaluated using an Patient Controlled Analgesia Pump

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Cesar Castello Branco, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No